CLINICAL TRIAL: NCT04459455
Title: Project HF-COVID: Evaluating Hyper-Brief, Online Materials During the COVID-19 Pandemic
Brief Title: Project H-COVID: Evaluating Hyper-Brief, Online Materials During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jessica Schleider, Assistant Professor of Psychology, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB2020-00204
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: We will use a between-subjects design; participants will be randomized to receive either the active Contain COVID Anxiety SSI or the placebo Remain COVID Free SSI
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This randomization of the order will occur using the randomizer within Qualtrics Survey Software, making the randomization process double-blind. To triple-blind our analysis process, the data will be downloaded from Qualtrics and the variable indicating what order the SSIs were presented in will be recoded before the primary analyses are conducted. Therefore, the primary analyses will be conducted without the knowledge of which condition is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contain COVID Anxiety SSI (Experimental): Participants first receive normalizing scientific information (including neuroscience findings) that help explain why increased anxiety during the COVID-19 is a typical response. They then read testimonials from three other people from the US who have applied a 3-step action plan for coping more effectively with their anxiety. The entire intervention takes approximately 8 minutes and is completely entirely within the Qualtrics survey platform.
  Interventions: Behavioral: Contain COVID Anxiety SSI
- Remain COVID Free SSI (Placebo Comparator): This placebo SSI was developed to mirror the structure of the Contain COVID Anxiety SSI, discuss COVID-19 related content, and do so without as many of the potential active ingredients of effective SSIs. Participants will receive scientific information about how soap kills the COVID-19 virus, but no neuroscience information related to behaviors or behavior change.
  Interventions: Behavioral: Remain COVID Free SSI

INTERVENTIONS:
Behavioral: Contain COVID Anxiety SSI — Participants first receive normalizing scientific information (including neuroscience findings) that help explain why increased anxiety during the COVID-19 is a typical response. They then read testimonials from three other people around the world who have applied a 3-step action plan for coping more effectively with their anxiety. The entire intervention takes approximately 8 minutes and is completely entirely within the Qualtrics survey platform.
  Arms: Contain COVID Anxiety SSI
Behavioral: Remain COVID Free SSI — This placebo SSI was developed to mirror the structure of the Contain COVID Anxiety SSI, discuss COVID-19 related content, and do so without as many of the potential active ingredients of effective SSIs. Participants will receive scientific information about how soap kills the COVID-19 virus, but no neuroscience information related to behaviors or behavior change.
  Arms: Remain COVID Free SSI

SUMMARY:
The goal of this study is to test whether an online, self-administered SSI designed to strengthen perceived control over anxiety in the context of the COVID-19 pandemic (Contain COVID Anxiety) increases perceived control over anxiety more than a placebo, hand-washing-plan SSI (Remain COVID Free) in a weighted-probability sample of the United States (N = 500).

DETAILED DESCRIPTION:
Elevations in state anxiety, when moderate and temporary, serve an adaptive function in pandemic contexts, facilitating health behaviors like self-protection and social distancing. However, for some people elevated state anxiety transitions to anxiety disorders, creating undue suffering and impairment. Nearly 33% of both Wuhan residents and Chinese citizens screened positive for generalized anxiety disorder during the COVID-19 pandemic, with uncontrollable, persistent COVID-19-related worries strongly predicting presence of GAD. Similarly, large surveys indicate that levels of anxiety symptoms are rising among United States citizens.

This finding aligns with a large body of literature indicating stronger perceived control over one's own anxiety buffers against a variety of anxiety disorders. Thus, in the context of COVID-19, there is a pressing need for materials that might strengthen perceived control over anxiety, thereby reducing risk for anxiety disorder onset. Ideally, such materials would (1) in no way undermine positive health behaviors, like social distancing, and (2) have capacity for broad-scale, immediate accessibility. Internet-based interventions may particularly valuable during the pandemic stage of COVID-19 due to the need for social distancing, and they have already scaled up to address needs in China. However, drop out from internet-based interventions can be up to 83% and intervention engagement is a frequent issue. Fortunately, single-session experiences (SSEs) can improve mental health related outcomes with similar effect sizes as multi-session therapies, and pilot data from our team suggests they can increase general perceived control (within-group dz = 0.70).

The goal of this project is to test a web-based platform where people can confidentially access and provide feedback on brief activities, called 'single-session experiences' (SSEs), which are about 8 minutes in length, entirely self-administered, and computer-based (Contain COVID Anxiety and Project Remain COVID Free). Previous activities following the same best practices as these experiences have been shown to be safe to complete; predicted significant reductions in psychological distress; and are entirely self-administered. We will recruit a weighted-probability sample of the United States through Prolific's online platform, N = 500. All data collected from the SSEs will be confidential, and the only identifiable information that will be recorded is the participants' Prolific ID to facilitate compensation, which will be deleted from the data after the compensation has been paid. Those that choose to complete the activities have the option to submit their advice to their peers and have it posted anonymously to the web-based platform. This will provide people with an option for an easily accessible activity designed to promote healthy coping skills and resilience in a welcoming environment through which they can learn with others and share experiences.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age is 18 years and older

Exclusion Criteria:

* Participant is younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Control Questionnaire (ACQ) from Baseline to Immediately Post-Intervention | Baseline, immediately post-intervention, 2-week follow-up
  ACQ is a 30-item questionnaire that measures an individual's level of agreement with a set of beliefs. Each item is scored on a scale from 0 (strongly disagree) to 5 (strongly agree) based on how much the statement is typical of the individual. The questionnaire measures domains of emotion control, threat control, and stress control, but only the emotion control scale (4 questions) will be used for the purposes of this study.
Change in Generalized Anxiety Disorder-7 (GAD-7) from Baseline to 2-week follow-up | Baseline, 2-week follow-up
  The GAD-7 asks participants to rate 7 statements based on how generally anxious they have felt over the past 2 weeks. Participants rate the 7 statements on a 4 point scale ranging from 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 21 with higher scores representing higher generalized anxiety.
Change in Activity Social Distancing Intentions - 3 item version (SOC-D) from Baseline to immediately post-intervention | Baseline, immediately post-intervention
  As validated measures for social distancing intentions do not yet exist, the 3 questions used in this measure are derived from the standardized item bank provided by the Center for Disease Control. The three questions ask participants to rate how long they believe others would be willing to engage in social distancing behaviors regarding large events, public spaces, and private gatherings. Participants rate the 3 statements on a 4 point scale ranging from 1 (Less than a Month) to 4 (4 months or more). Total score ranges from 4 to 12, with a higher score indicating greater levels of intention to socially distance.

SECONDARY OUTCOMES:
COVID-19 Related Questions | Baseline
  Derived from the CDC COVID-19 Community Survey Question Bank, participants will be asked to report whether they have been tested for COVID-19, tested positive for COVID-19, and displayed symptoms of COVID-19 in the past week. The questions also ask how the COVID-19 outbreak affected the participant in the past two weeks and if the children's schools are currently closed.
Inventory of Depression and Anxiety Symptoms (IDAS) | Baseline
  The IDAS is a screening tool for depression and panic disorder that asks people to rate how they have been feeling and acting in the past two weeks. Only the dysphoria subscale will be used; the subscale consists of 10 statements which the participants rate on a 1 (Not at all) to 5 (Extremely). Total score ranges from 10 to 50 for Dysphoria.
Self Hate Scale (SHS) | Baseline
  This brief measure asks participants to rate 7 statements measuring feelings of self-hatred on a 7-point Likert scale ranging from 1 (Not at all true for me) to 7 (Very true for me). Total score ranges from 7 to 49 with higher scores indicating higher levels of self hate.
Comprehension Questions | Immediately post-intervention
  Two multiple choice questions developed for the purpose of the study to serve as a quality check that ensures participants comprehended the core messages of both interventions.
Everyday Discrimination Scale-Short version | Baseline
  The 5-item measure assesses chronic and routine unfair treatment in daily life on a scale from 1 - 5, with a total score between 5 and 25
Perceived Changes in generalized anxiety symptoms | 2-week follow-up
  One question designed for use in this study. Participants rate their perceived changes in levels of generalized anxiety symptoms over 2 weeks from 1 (Much less anxiety) to 5 (much more anxiety)
Activity Hand Washing Intentions - 3 item version (WASH-I) | Baseline, immediately post-intervention
  This scale asks participants to rate 3 statements based on their intentions to engage in hand washing behaviors. Participants rate the 3 statements on a 7 point scale ranging from 1 (Strongly Agree) to 7 (Strongly Disagree). Total score ranges from 3 to 21, and will be reverse scored so a higher score indicates greater levels of intention to engage in recommended hand washing behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

REFERENCES:
- [Derived] Mullarkey M, Dobias M, Sung J, Ahuvia I, Shumake J, Beevers C, Schleider J. Web-Based Single Session Intervention for Perceived Control Over Anxiety During COVID-19: Randomized Controlled Trial. JMIR Ment Health. 2022 Apr 12;9(4):e33473. doi: 10.2196/33473. PMID 35230962